CLINICAL TRIAL: NCT00980070
Title: The Effectiveness of a Pediatric Lumbar Puncture Restraint Device
Acronym: SNOWBOARD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Angela Boettner, coordinator, University of Nebraska
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 329-09-FB
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Indication for Lumbar Puncture
Keywords: lumbar puncture positioning device
MeSH Terms: interventions — Spinal Puncture; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positioning Device (Experimental): use of positioning device
  Interventions: Device: Pediatric Restraint for Lumbar Puncture; Device: Lumbar Puncture Device
- Control (Active Comparator): institutional standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Pediatric Restraint for Lumbar Puncture — Restraint for children 1-90 days of age that allows physician to position pt for optimal lumbar puncture procedure.
  Arms: Positioning Device
Device: Lumbar Puncture Device — Lumbar Puncture positioner
  Other Names: Lumbar Puncture positioner
  Arms: Positioning Device
Other: Standard of Care — Lumbar Puncture positioner
  Arms: Control

SUMMARY:
This is a pilot study to evaluate a restraint device for lumbar punctures. Designed to help improve the restraint techniques for lumbar puncture, the restraint device will be compared to the current standard of manual physical restraint in neonatal and pediatric patients (age 1 day to 90 days of life). The investigators will study 30 subjects, with 20 randomized for the experimental device and 10 randomized for the "control" group, which is current standard of care. The investigators' primary outcomes will include time of procedure, red blood cells in the cerebrospinal fluid as well as physician satisfaction. Subjects will be eligible if they are 1-90 days of life, and their treating physician believes lumbar puncture is indicated. There is no follow-up once the lumbar puncture has been completed and the data has been obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 90 days of life
* Indication for lumbar puncture procedure as determined by the treating physician
* Informed Consent from the subject's legal guardian indicating their acceptance of a lumbar puncture for the work-up of sepsis
* Informed consent to enrolled in said protocol

Exclusion Criteria:

* No indication for lumbar puncture procedure as determined by treating physician

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of the lumbar puncture restraint board | one time use

SECONDARY OUTCOMES:
To evaluate the effect of the restraint board on the quality of the procedure (time of procedure, quality of specimen obtained, physician impression) | One time use

CONTACTS AND LOCATIONS:
Overall Officials: Edward Truemper, MD, Principal Investigator — UNMC
Locations (1):
- Childrens Hospital & Medical Center, Omaha, Nebraska, United States